CLINICAL TRIAL: NCT04733326
Title: Evaluation of Post-operative Pain and Expression of IL-8 Using Different Irrigate as Compared to Cryotherapy for Single Visit Endodontic Treatment in Teeth With Symptomatic Irreversible Pulpitis and Apical Periodontitis.Randomized Clinical Trial.
Brief Title: Evaluation of Post-operative Pain and Expression of IL-8 Using Ketolac or Cryoirrigation as a Final Flush in Single Visit Endodontic Treatment in Teeth With Symptomatic Irreversible Pulpitis and Apical Periodontitis.Randomized Clinical Trial.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yousra Khaled Mohamed Ezzat, BDS, MsC, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CairoU0
Record Dates: First submitted 2021-01-24; First posted 2021-02-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketorolac Tromethamine; Cryotherapy; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Participants presenting with symptomatic irreversible pulpits and apical periodontitis in their mandibular molars
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants didn't know to which group they are allocated and the outcome assessor received the data in an excel sheet
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cryothrapy (Experimental): 5 ml Saline at low temperature (2.5°C) will be used as intra-canal irrigantion during single visit endodontics treatment, to study the effect on reduction of post-operative pain and expression of IL-8.
  Interventions: Other: Cryotherapy
- Ketroloc tromethamine (Experimental): 2ml 30 mg Ketroloc tromethamine will be used as intra-canal irrigantion during single visit endodontics treatment, to study the effect on reduction of post-operative pain and expression of IL-8.
  Interventions: Drug: Ketorolac Tromethamine
- Saline at room temperature (Placebo Comparator): 30 ml Saline at room temperature will be used as intra-canal irrigantion during single visit endodontics treatment, to study the effect on reduction of post-operative pain and expression of IL-8.
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Ketorolac Tromethamine — final rinse with non-steriodal anti-inflammatory drug during single visit endodontic treatment in mandibular molar teeth with symptomatic irreversible pulpits and apical periodontitis
  Other Names: Ketolac
  Arms: Ketroloc tromethamine
Other: Cryotherapy — final rinse with cold saline during single visit endodontic treatment in mandibular molar teeth with symptomatic irreversible pulpits and apical periodontitis
  Other Names: Cold saline
  Arms: Cryothrapy
Other: Saline — final rinse with saline at room temperature during single visit endodontic treatment in mandibular molar teeth with symptomatic irreversible pulpits and apical periodontitis
  Arms: Saline at room temperature

SUMMARY:
To compare the effect of cryotherapy versus ketorolac tromethamine irrigating solutions used as a final flush in single visit endodontic treatment in mandibular molars, with symptomatic irreversible pulpitis and apical periodontitis on the:

* Intensity of post-operative pain in patients with symptomatic irreversible pulpitis
* Reduction of expression of Interleukin-8 (IL-8) post-instrumentation using ELISA
* The analgesic intake following endodontic treatment for post-operative pain relief.

DETAILED DESCRIPTION:
The main rationale of endodontic treatment is to eliminate micro-organisms from the infected root canal system by adequate chemo-mechanical debridement followed by a three-dimensional hermetic seal to provide a conductive environment for peri-radicular healing. However, Even with the utmost care in performing root canal therapy, it has been reported that the prevalence of post-operative pain after single visit endodontic treatment has been reported to be between 3 to 58%.

Non-steroidal anti-inflammatory drugs (NSAIDs) and Steroids have been advocated for control of post-operative pain following root canal treatment in teeth with symptomatic irreversible pulpitis. Ketorolac tromethamine, a potent NSAID that is over 400 times a selective inhibitor for COX-1 over COX-2 as compared to other drugs. In a recent study by (Evangelin et al 2019), assessing the influence of ketorolac tromethamine and dexamethasone when used as root canal irrigant on the expression of substance P and IL-8; showed that dexamethasone irrigation achieved the least post-operative pain and the least requirements for analgesics, whilst ketorolac tromethamine had better control on the expression of substance P and IL-8 as compared to dexamethasone.

Additionally, a more recent strategy for reduction of post-operative pain is cryotherapy. Such treatment modality is aimed to expose the body to very cold temperature, resulting in vasoconstriction and decreased permeability thus reducing the amount of fluid leaking into the peri-radicular tissues as exudate which commonly occur after chemo-mechanical preparation. Analgesia is closely related to the nerve conduction velocity of the nociceptive sensory nerve fibers. Thus, cooling induces analgesia by slowing the velocity of nerve conduction as well as decreasing the activation threshold of tissue nociceptors resulting in cold-induced neuropraxia. Thus the analgesic effect of cooling is produced by combination of decreased release of chemical mediators of pain and a slower propagation of neural pain signals.

In our study, ketorolac tromethamine, dexamethasone and cryotherapy are supposed to be used as root canal irrigants during root canal treatment to assess their effectiveness in reducing post-operative pain following single visit endodontic treatment in patients with symptomatic irreversible pulpitis, as well as their efficacy in reducing the expression of IL-8. Randomized clinical trials are the gold standard of interventional trials resulting in the highest level of evidence that contributes effectively in the clinical decision-making process as to the best intervention for the patient's condition providing the most effective clinical outcomes for the satisfaction of the patient. Thus the aim of the study is to compare the effect of using cryotherapy versus ketorolac tromethamine and dexamethasone irrigating solutions on the intensity of post-operative pain and reduction of expression of Interleukin-8(IL-8) post-instrumentation in patients with symptomatic irreversible pulpitis.

ELIGIBILITY:
Inclusion Criteria:

* - Medically free patients
* Age between 18-40 years old
* Males or females
* Participants able to understand Visual Analogue Scale (the pain chart diary) and sign the informed consent ( Appendix I,II).
* Mandibular permanent molar teeth:

  * Diagnosed clinically with symptomatic irreversible pulpitis associated with apical periodontitis.
  * Presence of spontaneous pain and sharp pain to cold tester (ethyl-chloride) that lingers after removal of the stimulus compared to the contra-lateral tooth
  * Tenderness to percussion with normal periapical radiographic appearance or slight widening of the lamina dura

Exclusion Criteria:

* - Participants allergic to NSAIDS
* Pregnant females
* Participants having significant systemic disorder
* If analgesics or antibiotics have been taken by the patient during the past 24 hours pre-operatively.
* Participants with psychological disturbances
* Participants with bruxism or clenching
* Participants having acute pain in more than one mandibular molar
* Participants with mandibular molar teeth showing:

  * Swelling or fistulous tract
  * Acute or chronic periapical abscess
  * Mobility greater than grade I
  * Periodontitis
  * Previous endodontic treatment or non-restorability

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Intensity of post-operative pain | 24 hours following endoodnitc treatment
  using the visual analogue scale

SECONDARY OUTCOMES:
IL-8 level | during root canal treatment
  using the ELISA
Analgesic intake | first 24 hours after completion of endodontic treatment
  counting the number of analgesic tablets taken after endodontic treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Cairo univresity, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No